CLINICAL TRIAL: NCT03565328
Title: Pilot Study to Evaluate the Effect of Nicotinamide Riboside on Skeletal Muscle Function in Heart Failure Subjects
Brief Title: The Effect of Nicotinamide Riboside on Skeletal Muscle Function in Heart Failure Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow/insufficient accrual and investigators have left the study.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 180107; 18-H-0107
Record Dates: First submitted 2018-06-20; First posted 2018-06-21 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: Mitochondrial bioenergetic dysfunction; Mitochondrial oxidative phosphorylation in skeletal muscles; Hyperacetylation of mitochondrial bioenergetic enzymes; NAD+ dependent sirtuin enzymes; NAD+/NADH ratio
MeSH Terms: conditions — Heart Failure | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotinamide Riboside in patients with stable heart failure (Experimental): Nicotinamide Riboside (NR) will be started at 500 mg daily (250 mg BID) then increased at two weekly intervals by 250 mg/dose (BID) (500 mg/day) to a final dose of 1000 mg PO BID (2000 mg/day) in patients with stable, systolic heart failure.
  Interventions: Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside (NR) will be started at 500 mg daily (250 mg BID) be increased at two weekly intervals by 250 mg/dose (BID) (500 mg/day) to a final dose of 1000mg PO BID (2000 mg/day).
  Other Names: Niagen; Nicotinamide Riboside (NR)

SUMMARY:
Background:

People are living longer and are more likely to survive a heart attack if they have one. Longer life expectancy is good but it also means more people get chronic heart failure over time. This is a condition in which the heart doesn't pump blood as well as it should. Treatment of chronic heart failure has not improved much in a few decades. Researchers want to see if giving a dietary supplement to people with heart failure can help their heart function. The supplement is nicotinamide riboside (NR).

Objective:

To study how NR affects skeletal muscle function in people with heart failure.

Eligibility:

Adults ages 18-70 with clinically stable systolic heart failure

Design:

Participants will be screened with a medical history and physical exam. They will answer demographic questions and review their current medical treatments. They will have blood and urine tests. They will have an echocardiogram. This uses sound waves to test heart function.

Participants will have 8 study visits over 16 weeks. At these visits, they will have some of the following:

Repeat of screening tests

Skin sample taken

Skeletal muscle exercise Nuclear magnetic resonance (NMR) spectroscopy. Muscles will be measured while participants do foot exercises.

Cardiopulmonary exercise testing. Participants may ride a stationary bike or walk on a treadmill. A facemask will analyze their breath. Heart and blood pressure measurements will be taken.

Participants will take the supplement in pill form each day for 12 weeks. Pill bottles will be checked at study visits.

Participants should not significantly change their activity levels during the study.

DETAILED DESCRIPTION:
As life expectancy increases and acute cardiac mortality decreases, the incidence of chronic heart failure (HF) continues to rise, and despite this, conceptual advances in the treatment of chronic heart failure have not increased substantially over last few decades. One intracellular component of heart failure progression is mitochondrial bioenergetic dysfunction. Although the mechanism underpinning this is not completely understood, recent metabolomics data demonstrated an incomplete flux of metabolites through oxidative phosphorylation (OX PHOS) in HF. In parallel, data has shown that hyperacetylation of mitochondrial bioenergetic enzymes, with the concomitant blunting of enzymatic activity is evident in HF. Putting these together, an emerging hypothesis implicates excessive acetylation of mitochondrial proteins with the subsequent blunting of bioenergetic enzyme function, as a mechanism underpinning incomplete flux through OX PHOS resulting in HF progression.

In parallel with cardiac bioenergetic deficiency chronic HF subjects display disrupted skeletal muscle OX PHOS, which is thought to contribute towards overall fatigue and reduced exercise tolerance. Interestingly exercise training in HF subjects improves skeletal muscle mitochondrial OX PHOS capacity and subject activity levels. Exercise training additionally increases activity of the mitochondrial regulatory deacetylase sirtuin enzymes SIRT1 and SIRT3, in parallel with improved skeletal muscle OX PHOS capacity. At the same time HF-associated disruption in skeletal muscle metabolic function activates skeletal muscle cytokine production. These inflammatory programs, in turn, are proposed to contribute towards impaired functional capacity in HF. Interestingly, and mirroring improved OX PHOS following exercise programs in HF studies, exercise training similarly reduces skeletal muscle inflammatory effects.

Biochemical and bioenergetic consequences of impaired mitochondrial OX PHOS leads to decreased NAD+ levels, which exacerbate mitochondrial dysfunction by inactivating the NAD+ dependent sirtuin enzymes. Experimental studies using NAD+ precursors to increase NAD+ production have been shown to normalize NADH/NAD+ ratios and activate Sirtuin enzymes, resulting in enhanced OX PHOS with beneficial effects in numerous systems including skeletal muscle and in the blunting of inflammation.

In this pilot study we will directly assess the effect of the NAD+ precursor, nicotinamide riboside (NR) on skeletal muscle mitochondrial OX PHOS in HF subjects using: skeletal muscle Nuclear magnetic resonance (NMR) spectroscopy assessment of the rate of high energy phosphate recovery in response to submaximal exercise; assessment of the effect of NR on functional capacity using cardiopulmonary exercise testing (CPET) to determine VO(2max) and anaerobic threshold; evaluation of the NR effect on serum metabolomics at rest and in response to CPET; and by measuring circulating cytokine levels pre- and post- NR administration. These studies would enable a more comprehensive assessment of the role for NR supplementation on skeletal muscle mitochondrial function in subjects with systolic HF

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women between the ages of 18 and 75 years with New York Heart Association (NYHA) Functional Classification Class II-III systolic heart failure ( Left Ventricular Ejection Fraction (LVEF) by standard echocardiography or radionuclide ventriculography of less than or equal to 45%) deemed to be non-ischemic or ischemic in origin.

Clinically stable (no cardiac procedures or hospitalizations for hospitalizations for cardiac causes, including HF, ischemia or arrhythmia) within the previous 3 months

Ability to undergo study procedures, including scheduled visits, blood draws, skeletal muscle exercise NMR spectroscopy and CPET testing

Willingness/ability to provide informed consent

Must be DEERS eligible to be enrolled in a research protocol at Walter Reed National Military Medical Center (WRNMMC).

EXCLUSION CRITERIA:

Heart failure with preserved ejection fraction (LVEF greater than 45%)

Change in heart failure medications due to deterioration of function with the exception of up- or down-titration of diuretic dose up to 100% of baseline dose.

Heart failure due to etiologies other than non-ischemic or ischemic. Examples of exclusionary heart failure etiologies include primary valvular disease, or infiltrative or inflammatory cardiomyopathies.

Cardiac surgery, percutaneous coronary intervention (PCI) or cardiac device implantation within the previous 3 months

Hospitalizations for cardiovascular causes, including heart failure, chest pain, stroke/TIA or arrhythmias within the previous 3 months

Inability to perform Study visits or procedures (e.g., physical inability to perform exercise testing)

Unwillingness/inability to provide informed consent

ALT greater than x3 upper limit of normal, hepatic insufficiency or active liver disease

Recent history of acute gout

Chronic renal insufficiency with creatinine greater than 2.5mg/dl

Pregnant (or likely to become pregnant) women

Significant co-morbidity likely to cause death in the 6 month follow-up period

Significant active history of substance abuse within the previous 5 years

Current participation in another drug study

History of intolerance to NR precursor compounds, including niacin or nicotinamide

MRI incompatible hardware including pacemakers or ICD s

Study adherence concerns

Individuals with diabetes type 1 and 2 who use insulin

Women of child-bearing potential unwilling to use contraception or unwilling to practice abstinence

Breastfeeding women unwilling to stop breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants signed informed consent: 1 subject completed the study; 1 subject failed the screening. Study was terminated due to lack of enrollment and precluded analysis of primary or secondary outcomes.
Period: Overall Study
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Enhancement of Mitochondrial Function in Skeletal Muscle
Description: Number of participants who had enhancement mitochondrial function in skeletal muscle Nuclear magnetic resonance (NMR) spectroscopy will be performed at baseline, at the end of the 12-week Nicotinamide Riboside (NR) supplementation period and repeated 4 weeks post-NR washout.
Time Frame: baseline-12 week-16 week
Population: 2 participants signed informed consent: 1 subject completed the study; 1 subject failed the screening. Study was terminated due to lack of enrollment and precluded analysis of primary or secondary outcomes.
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 0

2. Secondary Outcome: Measure the Effects of Nicotinamide Riboside (NR) on Oxidative Phosphorylation and Inflammation in Respective Subject Primary Skin Fibroblasts
Description: Measure the effects in participants of Nicotinamide Riboside (NR) on oxidative phosphorylation and inflammation in respective subject primary skin fibroblasts
Time Frame: Baseline, 12 week
Population: as for outcome 1
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Without Heart Failure Linked Inflammation
Description: To quantitative serum cytokine immunoassay profiling to assess whether Nicotinamide Riboside (NR) blunts heart failure (HF) linked inflammation
Time Frame: Baseline, 12 week
Population: as for outcome 1
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Experienced an Increased Rate of Oxidative Phosphorylation
Description: Serum quantitative metabolomic profiling, pre and post-cardiopulmonary exercise testing (CPET) to evaluate whether Nicotinamide Riboside (NR) increases the rate of oxidative phosphorylation
Time Frame: Baseline, 12 week
Population: as for outcome 1
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 0

5. Secondary Outcome: VO2 Max and Anaerobic Thresholds
Description: Analysis of VO2max and the anaerobic threshold will be measured.
Time Frame: Baseline, 12 week
Population: as for outcome 1
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Nicotinamide Riboside in Patients With Stable Heart Failure
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03565328/Prot_SAP_000.pdf